CLINICAL TRIAL: NCT05579548
Title: A Global, Multicenter Study to Assess Maternal, Fetal and Infant Outcomes of Exposure to Palynziq® (Pegvaliase) During Pregnancy and Breastfeeding
Acronym: PALomino
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Other Study IDs: 165-504
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonuria, Maternal
Keywords: Phase 4; Observational; Maternal; Pregnancy Outcomes; Exposure; Breastfeeding Outcomes
MeSH Terms: conditions — Phenylketonuria, Maternal | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women with PKU: This study will enroll pregnant women diagnosed with PKU who have been treated with pegvaliase from 2 weeks prior to LMP or at any time during pregnancy.
  Interventions: Drug: Pegvaliase

INTERVENTIONS:
Drug: Pegvaliase — Pregnant women exposed to pegvaliase within 2 weeks prior to LMP.

SUMMARY:
This is a Phase 4 observational study designed to assess the impact of Palynziq ® (pegvaliase) treatment in pregnant women with PKU and on their offspring who were exposed to pegvaliase at any time during pregnancy and breastfeeding.

DETAILED DESCRIPTION:
Women prescribed pegvaliase by their healthcare provider (HCP) who become pregnant during treatment may decide to participate in the study and enroll via a centralized call center model. Upon consent, data will be collected from the patient's HCP(s) retrospectively for at least 3 months prior to Last Menstrual Period (LMP). Data will be collected during pregnancy and throughout the infant's first year of life. Pegvaliase exposure will be recorded during pregnancy and breastfeeding including exposure during each trimester of pregnancy. Duration of individual subject participation will be up to approximately 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or a legally authorized representative) consent obtained prior to enrollment. Consent will be obtained in compliance with any country-specific regulations or requirements
* Confirmation of ongoing pregnancy. Subjects with unknown outcomes will be classified as prospective pregnancies; subjects who have undergone prenatal testing (eg, targeted ultrasound, amniocentesis) regardless of findings will be classified as retrospective pregnancies
* Diagnosed with PKU per local standard of care
* Documentation that the subject was treated with pegvaliase at any point starting from 2 weeks prior to the date of LMP
* Agrees to permit the Investigator (ie, CRP, CCA, PI) to contact the subject's HCPs (eg, PCP, PKU-treating physician, OB, nurse, midwife) and the infant's HCP (eg, pediatrician, neonatologist) for medical information

Exclusion Criteria:

• Currently participating in a BioMarin sponsored interventional study of any investigational product, device, or procedure

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only pregnant women with PKU who have been treated with Palynziq (pegvaliase) within 2 weeks of their last menstrual period are eligible.
Study Population: Pregnant women with PKU who have been treated with Palynziq (pegvaliase) within 2 weeks of their last menstrual period
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2032-10-04 (Estimated); Study Completion 2032-10-04 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome and infant development for women who have been treated with Palynziq (pegvaliase) within 2 weeks of their last menstrual period | 10 years
  To estimate the frequency of pregnancy outcomes (eg, spontaneous abortion, stillbirth, live birth, and termination) among subjects with PKU treated with pegvaliase during pregnancy and fetal/infant outcomes (all major congenital malformations [MCMs] and specifically microcephaly and congenital heart defects], FGR, small for gestational age [SGA], low birth weight, preterm birth, failure to thrive, and developmental delays) among their offspring exposed to pegvaliase during pregnancy.

SECONDARY OUTCOMES:
Pregnancy Outcomes | 10 years
  To compare the frequency of pregnancy outcomes (eg, spontaneous abortion, stillbirth, live birth, and termination) and fetal/infant outcomes (all MCMs and specifically microcephaly and congenital heart defects, FGR, SGA, low birth weight, preterm birth, failure to thrive, and developmental delays) among subjects with PKU treated with pegvaliase during pregnancy and their offspring to information on those same outcomes in non-pegvaliase exposed, pregnant women with PKU as described in reference literature
Pregnancy Outcomes | 10 years
  To examine differences in the frequency of pregnancy outcomes (eg, spontaneous abortion, stillbirth, live birth, and termination) and fetal/infant outcomes (all MCMs and specifically microcephaly and congenital heart defects, FGR, SGA, low birth weight, preterm birth, failure to thrive, and developmental delays) among subjects with PKU treated with pegvaliase during pregnancy and their offspring by maternal blood Phe levels
Serious Adverse Events | 10 years
  To estimate the frequency of serious adverse events (SAEs) other than CMs in infants exposed to pegvaliase during pregnancy through their first year of life
Maternal Pegvaliase use during breastfeeding | 10 years
  To estimate the frequency of selected outcomes in subjects with PKU treated with pegvaliase during breastfeeding (low milk supply) and their infants (failure to thrive and SAEs) through their first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- Syneos Health, Wilmington, North Carolina, United States
- Metabolics and Genetics in Calgary (MAGIC), Calgary, Canada
- Universitaetsklinikum Hamburg Eppendorf, Hamburg, Germany
- Ospedale San Paolo, Milan, Italy

REFERENCES:
- See also: Related Info — http://palomino-study.com/